CLINICAL TRIAL: NCT03141190
Title: Mindfulness Training to Improve Mental Health, Stress and Performance In Physicians
Brief Title: Mindful Mental Training for Surgeons to Enhance Resilience and Performance Under Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-19688
Record Dates: First submitted 2017-05-01; First posted 2017-05-05 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Burnout Syndrome; Surgery; Stress
Keywords: stress, surgery, mindfulness, feasibility
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Randomized, partially-blinded
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants do not know we are testing mindfulness only that they will be learning stress-reduction skills for surgeons
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Training for Surgeons (Experimental): Mindfulness-Based Stress Reduction (MBSR, as published elsewhere extensively) slightly modified by shortening the eight weekly classes to 2 hours each and the home practice requirement to 20 minutes. Taught by a veteran MBSR teacher with greater than 10,000 hours of personal practice and nearly 10 years of formal MBSR teaching experience.
  Interventions: Behavioral: Mindfulness Based Stress Reduction - modified
- The Mind of a Surgeon (Active Comparator): 8 weekly classes of 2 hours each with group reading and discussion of selected articles and stories about the ethos and experience of becoming a surgeon. Designed and administered by a surgical faculty member with extensive experience in surgical education and scholarly work in the area of the 'surgical personality'.
  Interventions: Behavioral: Active listening and reading

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction - modified — already described
  Other Names: MBSR
  Arms: Mental Training for Surgeons
Behavioral: Active listening and reading — group reading, listening and discussion of articles pertaining to the development and experience of the surgical personality
  Arms: The Mind of a Surgeon

SUMMARY:
Background:

Burnout and overwhelming stress are growing issues among surgeons and are associated with mental illness, attrition and diminished patient care. Among surgical trainees, burnout and distress are alarmingly prevalent but high inherent mindfulness has been shown to decrease the risk of depression, suicidal ideation, burnout and overwhelming stress by more than 75%. In other high-stress populations formal mindfulness training has been shown to improve mental health and buffer overwhelming stress and yet this approach has not been tried in surgery.

The aim of this study is to evaluate feasibility and acceptability of modified mindfulness-based stress reduction (MBSR) training among PGY-1 surgery residents and to obtain initial evidence of efficacy in regard to well-being and performance.

Design: A pilot randomized clinical trial of modified MBSR versus an active control.

Setting: Residency training program, tertiary academic medical center.

Participants: PGY-1 surgery residents.

Intervention:

Weekly two-hour modified MBSR classes (compared to an active control) and 20 minutes of suggested daily home practice over an eight-week period.

Main Outcomes and Measures:

Primary outcome is feasibility, assessed along six domains (demand, implementation, practicality, acceptability, adaptation and integration), using focus groups, interviews, surveys, attendance, daily practice time and subjective self-report of experience.

Secondary outcomes include perceived stress, mindfulness and executive function (specifically working memory capacity), followed by psychosocial well-being (burnout, depression, resilience), performance (motor skills testing) and functional brain scans focused on areas associated with reappraisal as a surrogate for emotional control.

This study seeks to demonstrate the feasibility of mindfulness training in surgery PGY-1s while simultaneously providing preliminary quantitative data on the effects of mindfulness training in a randomized, controlled setting. Data will inform modifications to the MBSR curriculum that enhance feasibility and inform sample size calculations for subsequent, adequately-powered RCTs which will likely need to be multi-center trials.

Results could potentially impact formal medical training, the mental health of providers at every level, and the overall quality of patient care.

DETAILED DESCRIPTION:
Mounting evidence shows that burnout, a critical metric for dissatisfaction and distress, is a growing problem within medicine. Burnout is a syndrome associated with worse physician performance, patient outcomes, and hospital economics.The quadruple aim of healthcare underscores that physician fulfillment is a critical part of any sustainable reform and appropriately frames physician burnout and fulfillment as issues that impact everyone, not just individual providers.

Burnout is believed to arise from a mismatch between expectations and reality, with more than half of practicing physicians and trainees reported to suffer from this problem. Among general surgery residents, the prevalence of burnout is estimated at 69% and dramatically increases the odds of both overwhelming stress and distress symptoms. The relationship between overwhelming stress and burnout is particularly concerning because extensive evidence links overwhelming stress to detrimental effects on learning, memory, decision-making, and performance.

A recent meta-analysis suggests that stress management/mindfulness interventions are particularly effective at addressing burnout on the individual level. Small cohort studies and controlled trials have shown mindfulness-based interventions to be effective at reducing stress and burnout in medical students, primary care physicians, internists, and other healthcare providers.

In general surgery trainees, inherent mindfulness tendencies (shown to increase following mindfulness training), decrease the risk of burnout, overwhelming stress, and distress symptoms by 75% or more. This suggests that mindfulness tendencies may already be used, albeit unconsciously, to cope within the high-stress culture of surgery. Indeed, isolated studies of performance strategies that involve emotional regulation, and focused attention (qualities shared with mindfulness training) have also demonstrated improvements in surgeons' technical performance and perceived stress.

Mindfulness meditation training involves the cultivation of moment-to-moment awareness of thoughts, emotions and sensations (also known as interoception), the development of non-reactivity in response to stimuli (also known as emotional regulation), and the enhancement of perspective-taking regarding oneself and others. The most scientifically studied form of mindfulness training is the secular Mindfulness-Based Stress Reduction (MBSR) developed by Jon Kabat-Zinn in the 1970s. MBSR is formally trained through an eight-week codified curriculum and has been shown to decrease stress and burnout, protect executive function, and enhance performance in multiple high-stress populations.

In spite of such evidence, mindfulness training among surgeons has only occasionally been suggested or informally pursued, partly due to a disconnect between the indefatigable stoicism of surgery and mindfulness, which is often perceived as relaxation rather than a skill to enhance resilience. Moreover, the time pressures of surgical training make additional responsibilities and new curricula seem impossible.

In fact, the global effects of mindfulness training, as opposed to other interventions that target a single outcome, may prove to be its biggest asset. Individuals don't manifest the effects of overwhelming stress and burnout in identical ways, making an up-stream intervention with myriad downstream effects the most efficient method for intervening on large, diverse populations. Moreover, while other forms of skills training or mental health interventions require recurrent time away from work, mindfulness training involves an initial investment of time but then can be strengthened through practice in everyday settings - within the daily life, not separate from it.

To systematically examine the feasibility of formal mindfulness training during surgery internship at a tertiary academic center, we undertook the "Mindful Surgeon" pilot study. Our secondary goal is to gather preliminary evidence of efficacy, to guide future design of a scalable, adequately powered trial.

ELIGIBILITY:
Inclusion Criteria:

* UCSF surgical interns entering training. Do not meet exclusion criteria.

Exclusion Criteria:

* Current personal mindfulness practice, medications with CNS effects, lifetime history of a mental disorder, acute or chronic immune or inflammatory disorders, pregnancy, breast-feeding or implanted MRI-incompatible metal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Stress | baseline, 8wks (post-intervention),12-month follow-up
  Cohen's Perceived Stress Scale (PSS)

SECONDARY OUTCOMES:
Change in Executive Function | baseline, 8wks (post-intervention),12-month follow-up
  Executive function as assessed via working memory capacity, cognitive control and executive composite components of the NIH EXAMINER battery.

OTHER OUTCOMES:
Change in Motor skills | baseline, 8wks (post-intervention),12-month follow-up
  Performance as assessed by the Fundamentals of Laparoscopic Surgery (FLS) modules
Change in Functional neuroanatomic changes | baseline, 8wks (post-intervention),12-month follow-up
  Functional changes in areas associated with reappraisal/emotional regulation (amygdala, hippocampus, reward circuitry, appraisal pathway) as evidenced by fMRI BOLD and DTI brain scans analyzed by whole brain and a prior region of interest approaches.
Change in Psychological well-being | baseline, 8wks (post-intervention),12-month follow-up
  burnout (Maslach burnout inventory), depression (PHQ-9), resilience (ER89), Grit (GRIT-S), mindfulness (CAMS-R)

CONTACTS AND LOCATIONS:
Overall Officials: Carter Lebares, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shanafelt TD, Hasan O, Dyrbye LN, Sinsky C, Satele D, Sloan J, West CP. Changes in Burnout and Satisfaction With Work-Life Balance in Physicians and the General US Working Population Between 2011 and 2014. Mayo Clin Proc. 2015 Dec;90(12):1600-13. doi: 10.1016/j.mayocp.2015.08.023. PMID 26653297
- [Background] Shanafelt TD, Balch CM, Bechamps G, Russell T, Dyrbye L, Satele D, Collicott P, Novotny PJ, Sloan J, Freischlag J. Burnout and medical errors among American surgeons. Ann Surg. 2010 Jun;251(6):995-1000. doi: 10.1097/SLA.0b013e3181bfdab3. PMID 19934755
- [Background] Scheepers RA, Boerebach BC, Arah OA, Heineman MJ, Lombarts KM. A Systematic Review of the Impact of Physicians' Occupational Well-Being on the Quality of Patient Care. Int J Behav Med. 2015 Dec;22(6):683-98. doi: 10.1007/s12529-015-9473-3. PMID 25733349
- [Background] Haas JS, Cook EF, Puopolo AL, Burstin HR, Cleary PD, Brennan TA. Is the professional satisfaction of general internists associated with patient satisfaction? J Gen Intern Med. 2000 Feb;15(2):122-8. doi: 10.1046/j.1525-1497.2000.02219.x. PMID 10672116
- [Background] DiMatteo MR, Sherbourne CD, Hays RD, Ordway L, Kravitz RL, McGlynn EA, Kaplan S, Rogers WH. Physicians' characteristics influence patients' adherence to medical treatment: results from the Medical Outcomes Study. Health Psychol. 1993 Mar;12(2):93-102. doi: 10.1037/0278-6133.12.2.93. PMID 8500445
- [Background] Del Canale S, Louis DZ, Maio V, Wang X, Rossi G, Hojat M, Gonnella JS. The relationship between physician empathy and disease complications: an empirical study of primary care physicians and their diabetic patients in Parma, Italy. Acad Med. 2012 Sep;87(9):1243-9. doi: 10.1097/ACM.0b013e3182628fbf. PMID 22836852
- [Background] Sinsky CA, Dyrbye LN, West CP, Satele D, Tutty M, Shanafelt TD. Professional Satisfaction and the Career Plans of US Physicians. Mayo Clin Proc. 2017 Nov;92(11):1625-1635. doi: 10.1016/j.mayocp.2017.08.017. Epub 2017 Nov 1. PMID 29101932
- [Background] Dyrbye LN, Trockel M, Frank E, Olson K, Linzer M, Lemaire J, Swensen S, Shanafelt T, Sinsky CA. Development of a Research Agenda to Identify Evidence-Based Strategies to Improve Physician Wellness and Reduce Burnout. Ann Intern Med. 2017 May 16;166(10):743-744. doi: 10.7326/M16-2956. Epub 2017 Apr 18. No abstract available. PMID 28418518
- [Background] Bodenheimer T, Sinsky C. From triple to quadruple aim: care of the patient requires care of the provider. Ann Fam Med. 2014 Nov-Dec;12(6):573-6. doi: 10.1370/afm.1713. PMID 25384822
- [Background] Campbell J, Prochazka AV, Yamashita T, Gopal R. Predictors of persistent burnout in internal medicine residents: a prospective cohort study. Acad Med. 2010 Oct;85(10):1630-4. doi: 10.1097/ACM.0b013e3181f0c4e7. PMID 20881685
- [Background] Center C, Davis M, Detre T, Ford DE, Hansbrough W, Hendin H, Laszlo J, Litts DA, Mann J, Mansky PA, Michels R, Miles SH, Proujansky R, Reynolds CF 3rd, Silverman MM. Confronting depression and suicide in physicians: a consensus statement. JAMA. 2003 Jun 18;289(23):3161-6. doi: 10.1001/jama.289.23.3161. PMID 12813122
- [Background] Karlamangla AS, Singer BH, McEwen BS, Rowe JW, Seeman TE. Allostatic load as a predictor of functional decline. MacArthur studies of successful aging. J Clin Epidemiol. 2002 Jul;55(7):696-710. doi: 10.1016/s0895-4356(02)00399-2. PMID 12160918
- [Background] Arora S, Sevdalis N, Aggarwal R, Sirimanna P, Darzi A, Kneebone R. Stress impairs psychomotor performance in novice laparoscopic surgeons. Surg Endosc. 2010 Oct;24(10):2588-93. doi: 10.1007/s00464-010-1013-2. Epub 2010 Mar 31. PMID 20354878
- [Background] Wetzel CM, Kneebone RL, Woloshynowych M, Nestel D, Moorthy K, Kidd J, Darzi A. The effects of stress on surgical performance. Am J Surg. 2006 Jan;191(1):5-10. doi: 10.1016/j.amjsurg.2005.08.034. PMID 16399098
- [Background] Jha AP, Stanley EA, Kiyonaga A, Wong L, Gelfand L. Examining the protective effects of mindfulness training on working memory capacity and affective experience. Emotion. 2010 Feb;10(1):54-64. doi: 10.1037/a0018438. PMID 20141302
- [Background] Seppala EM, Nitschke JB, Tudorascu DL, Hayes A, Goldstein MR, Nguyen DT, Perlman D, Davidson RJ. Breathing-based meditation decreases posttraumatic stress disorder symptoms in U.S. military veterans: a randomized controlled longitudinal study. J Trauma Stress. 2014 Aug;27(4):397-405. doi: 10.1002/jts.21936. PMID 25158633
- [Background] Amutio A, Martinez-Taboada C, Delgado LC, Hermosilla D, Mozaz MJ. Acceptability and Effectiveness of a Long-Term Educational Intervention to Reduce Physicians' Stress-Related Conditions. J Contin Educ Health Prof. 2015 Fall;35(4):255-60. doi: 10.1097/CEH.0000000000000002. PMID 26953856
- [Background] Johnson DC, Thom NJ, Stanley EA, Haase L, Simmons AN, Shih PA, Thompson WK, Potterat EG, Minor TR, Paulus MP. Modifying resilience mechanisms in at-risk individuals: a controlled study of mindfulness training in Marines preparing for deployment. Am J Psychiatry. 2014 Aug;171(8):844-53. doi: 10.1176/appi.ajp.2014.13040502. PMID 24832476
- [Background] Lebares CC, Guvva EV, Ascher NL, O'Sullivan PS, Harris HW, Epel ES. Burnout and Stress Among US Surgery Residents: Psychological Distress and Resilience. J Am Coll Surg. 2018 Jan;226(1):80-90. doi: 10.1016/j.jamcollsurg.2017.10.010. Epub 2017 Oct 26. PMID 29107117
- [Background] Wager TD, Davidson ML, Hughes BL, Lindquist MA, Ochsner KN. Prefrontal-subcortical pathways mediating successful emotion regulation. Neuron. 2008 Sep 25;59(6):1037-50. doi: 10.1016/j.neuron.2008.09.006. PMID 18817740
- [Background] Krasner MS, Epstein RM, Beckman H, Suchman AL, Chapman B, Mooney CJ, Quill TE. Association of an educational program in mindful communication with burnout, empathy, and attitudes among primary care physicians. JAMA. 2009 Sep 23;302(12):1284-93. doi: 10.1001/jama.2009.1384. PMID 19773563
- [Result] Lebares CC, Coaston TN, Delucchi KL, Guvva EV, Shen WT, Staffaroni AM, Kramer JH, Epel ES, Hecht FM, Ascher NL, Harris HW, Cole SW. Enhanced Stress Resilience Training in Surgeons: Iterative Adaptation and Biopsychosocial Effects in 2 Small Randomized Trials. Ann Surg. 2021 Mar 1;273(3):424-432. doi: 10.1097/SLA.0000000000004145. PMID 32773637
- [Result] Lebares CC, Hershberger AO, Guvva EV, Desai A, Mitchell J, Shen W, Reilly LM, Delucchi KL, O'Sullivan PS, Ascher NL, Harris HW. Feasibility of Formal Mindfulness-Based Stress-Resilience Training Among Surgery Interns: A Randomized Clinical Trial. JAMA Surg. 2018 Oct 1;153(10):e182734. doi: 10.1001/jamasurg.2018.2734. Epub 2018 Oct 17. PMID 30167655
- [Result] Lebares CC, Guvva EV, Olaru M, Sugrue LP, Staffaroni AM, Delucchi KL, Kramer JH, Ascher NL, Harris HW. Efficacy of Mindfulness-Based Cognitive Training in Surgery: Additional Analysis of the Mindful Surgeon Pilot Randomized Clinical Trial. JAMA Netw Open. 2019 May 3;2(5):e194108. doi: 10.1001/jamanetworkopen.2019.4108. PMID 31125095
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860